CLINICAL TRIAL: NCT03504202
Title: Effect of Trimetazidine on the Improvement of Coronary Microvascular Dysfunction in Patients With INOCA(Ischemia and no Obstructive Coronary Artery Disease)
Acronym: T-MICRO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Ya-Wei Xu, The chief director of department of cardiology, Shanghai 10th People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T-MICRO01
Record Dates: First submitted 2018-04-11; First posted 2018-04-20 (Actual); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Patients With INOCA(Ischemia and no Obstructive Coronary Artery Disease) Who Have Coronary Microvascular Dysfunction
MeSH Terms: interventions — Trimetazidine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Trimetazidine (Experimental)
  Interventions: Drug: Trimetazidine

INTERVENTIONS:
Drug: Trimetazidine — After enrollment, experimental group will receive Trimetazidine(35mg tid) for six months .

SUMMARY:
This is a prospective study which aims to explore the effect of Trimetazidine on the improvement of coronary microvascular dysfunction in patients with INOCA (ischemia and no obstructive coronary artery disease). Enrolled patients will be assessed SAQ(Seattle Angina Score), Canadian Angina Grade(Canadian Cardiovascular Society, CCS), Six-Minute Walk Test, CFR(coronary flow reserve) .CFR inspection with D-SPECT and pressure guide wire.Patients will receive six months Trimetazidine(35mg tid) after enrollment. And their SAQ (Seattle Angina Score), Canadian Angina Grade(Canadian Cardiovascular Society, CCS), Six-Minute Walk Test, CFR will be followed up.

ELIGIBILITY:
Inclusion Criteria:

* age≥18 years
* Typical angina symptoms
* Coronary angiography or coronary computed tomography examination showed no significant epicardial coronary artery stenosis (<20%)
* Never used trimetazidine
* The CFR measured by the pressure guide wire is less than 2.0
* agree to participant the study and sign informed written consent
* available for six months follow up

Exclusion Criteria:

* Severe liver and kidney disease
* Contraindications of Trimetazidine
* Use of CYP3A inhibitors, such as diltiazem, verapamil, and other drugs that may affect CFR measurements
* QT interval extension
* Atrial fibrillation or left bundle branch block
* Left ventricular systolic dysfunction (EF <55%)
* Coronary artery fistula
* Myocardial bridge
* Non-cardiogenic chest pain and other heart diseases
* Severe heart valve disease
* Diabetes
* Recent ACS( Acute coronary syndrome)
* Pregnancy
* Failed to complete inspection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-03-01 (Estimated); Primary Completion 2020-04-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
Coronary flow reserve (CFR) improves | six months

SECONDARY OUTCOMES:
Seattle angina score or Canadian angina grade drops | six months
Six-minute walking experiment improves | six months